CLINICAL TRIAL: NCT00281333
Title: The Influence of "Karate" on Bleeding in Hemophilic Patients.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: logistics
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sheba Medical Center, Sheba Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SHEBA-02-2708-UM-CTIL
Record Dates: First submitted 2006-01-23; First posted 2006-01-24 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: "Karate" exercises and strengthening exercises

SUMMARY:
Hemophilia patients tend to lower their physical activity level due to the fear of increasing bleeding episodes. Although recent literature has shown that with routine muscle strengthening and physical activity, the frequency and duration of bleeds was reduced. Our study has built a routine of strength training exercises and karate training. The study is built in two stages, each stage being three months. The participants fill out a bleeding diary that includes information from the previous six months. It includes place of bleed, duration, pain level, spontaneous or traumatic bleed, factor replacement and joint limitation. Before the exercise, the participants are tested for muscle strength and endurance. The bleeding diary will be filled out following the first three months and the second phase as will the muscle strength and endurance. We are hoping to see a drastic reduction of bleeding episodes occurring especially from spontaneous bleeds.

DETAILED DESCRIPTION:
none - Hemophilia patients tend to lower their physical activity level due to the fear of increasing bleeding episodes. Although recent literature has shown that with routine muscle strengthening and physical activity, the frequency and duration of bleeds was reduced. Our study has built a routine of strength training exercises and karate training. The study is built in two stages, each stage being three months. The participants fill out a bleeding diary that includes information from the previous six months. It includes place of bleed, duration, pain level, spontaneous or traumatic bleed, factor replacement and joint limitation. Before the exercise, the participants are tested for muscle strength and endurance. The bleeding diary will be filled out following the first three months and the second phase as will the muscle strength and endurance. We are hoping to see a drastic reduction of bleeding episodes occurring especially from spontaneous bleeds.

ELIGIBILITY:
Inclusion Criteria:

* Severe Hemophilia.

Exclusion Criteria:

* No Inhibitors.

Ages: 11 Years to 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uri Martinowitz, M.D., Principal Investigator — Sheba Medical Center